CLINICAL TRIAL: NCT03198533
Title: Evaluation of Triathlon - A New Total Knee Prosthesis System - Triathlon PA vs. Triathlon Pressfit
Acronym: TriathlonRSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-S-015 Triathlon RSA _3
Record Dates: First submitted 2017-05-09; First posted 2017-06-26 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee; Arthrosis; Implant
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triathlon PA (Active Comparator): Triathlon PA (HA-surface) versus Triathlon Pressfit design: The goal with the un-cemented technique is to reach a full integration between the bone and the prosthesis. During the last years the usage of prosthesis with hydroxyapatite surface within tooth-, mandibular-surgery, hips- and knee-joints, have increased significantly. It has been shown that a thin layer of hydroxyapatite stimulates the anchorage of the implant. The goal with this sub study is to compare the stability of the fixation when using two different types of Triathlon un-cemented prosthesis designs. PA (HA-surface) versus Pressfit.
  Interventions: Device: Triathlon PA
- Triathlon Pressfit (Active Comparator): Triathlon PA (HA-surface) versus Triathlon Pressfit design: The goal with the un-cemented technique is to reach a full integration between the bone and the prosthesis. During the last years the usage of prosthesis with hydroxyapatite surface within tooth-, mandibular-surgery, hips- and knee-joints, have increased significantly. It has been shown that a thin layer of hydroxyapatite stimulates the anchorage of the implant. The goal with this sub study is to compare the stability of the fixation when using two different types of Triathlon un-cemented prosthesis designs. PA (HA-surface) versus Pressfit.
  Interventions: Device: Triathlon Pressfit

INTERVENTIONS:
Device: Triathlon PA — Implantation of Knee Prosthesis
  Arms: Triathlon PA
Device: Triathlon Pressfit — Implantation of Knee Prosthesis
  Arms: Triathlon Pressfit

SUMMARY:
The objective is to investigate the Clinical, Radiographic, Roentgen Stereophotogrammetric behaviour and patient outcome when using the Triathlon total knee prosthesis in a prospective randomized clinical trial.

DETAILED DESCRIPTION:
The objective is to investigate the Clinical, Radiographic, Roentgen Stereophotogrammetric behaviour and patient outcome when using the Triathlon total knee prosthesis in a prospective randomized clinical trial.

The evaluation is carried out by a prospective randomised RSA-study with Triathlon PA vs. Triathlon Pressfit

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering exclusively from OA, Stage II-V [Ahlbäck, 1968 391] will be operated.
2. Patients requiring knee prosthesis, suitable for the use of Duracon and Triathlon knee system
3. Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographical evaluations and the prescribed rehabilitation.
4. Patients who signed the Ethics Committee approved Informed Consent Form prior to surgery.

Exclusion Criteria:

1. Previous major knee surgery
2. Other significant disabling problems from the muscular-skeletal system than in the knees
3. Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2: BMI above 35).
4. Patients with active or suspected infection.
5. Patients with malignancy - active malignancy.
6. Patients with severe osteoporosis, Paget's disease, renal osteodystrophy.
7. Patients immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
8. The patient has a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
9. Female patients planning a pregnancy during the course of the study.
10. Patients with systemic or metabolic disorders leading to progressive bone deterioration.
11. Patients, who as judged by the surgeon, are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
12. Patients with other severe concurrent joint involvements, which can affect their outcome.
13. Patients with other concurrent illnesses, which are likely to affect their outcome such as sickle cell anaemia, systemic lupus erythematosus or renal disease requiring dialysis.
14. Patients under the protection of law (e.g. guardianship).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07-10 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Roentgen Stereophotogrammetric Analysis (RSA) | 10 years follow-up
  Assessment of fixation and stability of the Triathlon total knee prosthesis by Roentgen Assessment of fixation and stability of the Triathlon total knee prosthesis by RSA as a predictor of late mechanical loosening.

SECONDARY OUTCOMES:
Investigation of clinical performance and patient outcome with the Knee Society Score (KSS) | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Investigation of clinical performance and patient outcome with the Knee Injury and Osteoarthritis Outcome Score (KOOS) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  KOOS consists of 5 subscales: Pain, other symptoms, function in daily living , function in sport and recreation and knee related quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms).
Investigation of clinical performance and patient outcome with EuroQuol-5 dimension (EQ-5D) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
Investigation of patient outcome with radiographic analysis | 3 months, 1, 2, 5, 7 and 10 years
  Plain radiographs will be obtained for assessment of fixation of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Sören Toksvig-Larsen, MD, Principal Investigator — Skånevård Kryh Division Kirurgi och Ortopedkliniken Hässleholm
Locations (1):
- Skånevård Kryh Division Kirurgi och Ortopedkliniken Hässleholm, Hässleholm, Skåne County, Sweden